CLINICAL TRIAL: NCT02321813
Title: Direct Improvement of Quality of Life Using a Tailored Pathway With Quality of Life Diagnosis and Therapy: Protocol of a Randomised Clinical Trial in Colorectal Cancer Patients
Brief Title: Direct Improvement of Quality of Life Using a Tailored Pathway With Quality of Life Diagnosis and Therapy: Randomised Trial in Colorectal Cancer Patients
Acronym: DIQOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tumor Center Regensburg (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Ass. Prof. Dr. Monika Klinkhammer-Schalke, PD Dr.med. Monika Klinkhammer-Schalke, Tumor Center Regensburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TUZ-QL-CRC-14; 01GY1339 (Other Grant/Funding Number: German Federal Ministry of Education and Research)
Record Dates: First submitted 2014-12-11; First posted 2014-12-22 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Quality of Life; Colorectal Neoplasms
Keywords: quality of life; colorectal cancer; definitive RCT; complex intervention
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention group (Experimental): In the quality of life pathway results of the quality of life (QoL) measure are transferred to a QoL-profile. Three experts with various professional background use the individual patient's QoL-profile and clinical and sociodemographic information in order to generate a QoL-report including therapy recommendation which is sent to the coordinating practitioner. Specific therapeutic options for the treatment of diseased QoL have been identified: pain therapy, psychotherapy, social support, nutrition counseling, stoma care, physiotherapy, fitness. To provide continuous medical education, quality circles for each therapy option haven been founded. Coordinating practitioners receive a list with addresses of all quality circle members.
  Interventions: Behavioral: quality of life pathway
- control group (Placebo Comparator): In control group QoL is also measured but the coordinating practitioner neither receives a QoL-profile nor a QoL-report.
  Interventions: Other: placebo control

INTERVENTIONS:
Behavioral: quality of life pathway — Quality of life measurement, diagnosis and tailored therapy (pain therapy, psychotherapy, social support, nutrition, stoma care, physiotherapy, fitness)
  Arms: intervention group
Other: placebo control — Quality of life measurement
  Arms: control group

SUMMARY:
The purpose of the study is to determine whether a quality of life pathway with defined diagnostic and therapeutic options improves quality of life in colorectal cancer patients during follow-up.

DETAILED DESCRIPTION:
There is a growing interest in using quality of life (QoL) data not only as relevant endpoint in clinical trials on cancer patients, but also in routine practice in order to improve patients' health during treatment. The investigators designed, implemented and evaluated an integrated quality of life diagnosis and therapy pathway (QoL pathway) for breast cancer patients (Klinkhammer-Schalke et al, 2008; 2012), guided by the UK Medical Research Council framework for developing and testing complex interventions. It could be demonstrated in a routine setting that breast cancer patients showed a benefit from tailored QoL diagnosis and therapy (Klinkhammer-Schalke et al, 2012).

But there is also requirement for managing QoL deficits of patients with other cancers and to replicate findings of the previous trial. To achieve this aim, the QoL pathway has been modified for colorectal cancer patients. The Tumor Center Regensburg provides the infrastructure of the present project (quality circles, project groups).

This is a two-arm randomised clinical trial with one intervention group and one control group. Patients' QoL is assessed with the EORTC QLQ-C30 and QLQ-CR29 at 0, 3, 6, 12, and 18 months after surgery.

In intervention group results of the QoL-measure are transferred to a QoL-profile including 13 dimensions on scales of 0-100 (cutoff for "diseased QoL <50). Three experts with varying professional background use the individual patient's QoL-profile and clinical and sociodemographic information in order to generate a QoL-report including therapy recommendation which is sent to the coordinating practitioner. Specific therapeutic options for the treatment of diseased QoL have been identified: pain therapy, psychotherapy, social support, nutrition counseling, stoma care, physiotherapy, fitness. To provide continuous medical education, quality circles for each therapy option have been founded. Coordinating practitioners receive a list with addresses of all quality circle members.

In control group QoL is also measured but the coordinating practitioner neither receives a QoL-profile nor a QoL-report.

The investigators expect that patients in the intervention group will experience a lower number of QoL-deficits (QoL < 50 points) in the first year after surgery compared with patients in the control group

ELIGIBILITY:
Inclusion Criteria:

* primary colorectal cancer
* operated in one of four participating certified cancer centres for colorectal cancer (Krankenhaus Barmherzige Brüder, Department of Surgery, Regensburg; Germany; Caritas-Krankenhaus St. Josef, Department of Surgery, Regensburg; Germany; Klinikum Neumarkt., Department of Surgery, Neumarkt; Germany; Klinikum St. Elisabeth Straubing, Department of Surgery, Straubing, Germany), documented in a population-based cancer registry (Tumor Center Regensburg e.V.)
* informed consent.

Exclusion Criteria:

* coordinating practitioner not implemented
* patient from district outside the study region (rural districts Regensburg, Neumarkt, Straubing, Straubing-Bogen, Kelheim, Schwandorf)
* patient unable to fill out the questionnaire for physical, psychological or language reasons (including dementia)
* age under 18 years
* pregnancy
* QoL clinician unavailable
* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2014-01; Primary Completion 2016-11 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
proportion of patients in both groups with diseased quality of life (<50 points in at least one dimension) | 1 year after the date of primary surgery for colorectal cancer

SECONDARY OUTCOMES:
rates of patients with diseased quality of life in each dimension of the profile | 0 (0-2 days before clinical discharge), 3, 6, 12, and 18 months after primary surgery for colorectal cancer

CONTACTS AND LOCATIONS:
Overall Officials: Monika Klinkhammer-Schalke, MD, Ass. Prof., Study Chair — Tumor Center Regensburg e.V., An-Institute of the University of Regensburg, Germany; Michael Koller, Ph.D., Prof., Principal Investigator — Center for Clinical Trials, University Regensburg, Germany; Wilfried Lorenz, MD, Prof. Ɨ, Principal Investigator — Tumor Center Regensburg e.V., An-Institute of the University of Regensburg, Germany; Ferdinand Hofstädter, MD, Prof., Principal Investigator — Johannes Kepler University Linz, Medical Faculty, Austria; Jeremy C Wyatt, MD, Prof., Principal Investigator — Leeds Institute of Health Sciences, University of Leeds, UK
Locations (1):
- Tumor Center Regensburg e.V., An-Institute of the University of Regensburg, Regensburg, Bavaria, Germany

REFERENCES:
- [Background] Klinkhammer-Schalke M, Koller M, Steinger B, Ehret C, Ernst B, Wyatt JC, Hofstadter F, Lorenz W; Regensburg QoL Study Group. Direct improvement of quality of life using a tailored quality of life diagnosis and therapy pathway: randomised trial in 200 women with breast cancer. Br J Cancer. 2012 Feb 28;106(5):826-38. doi: 10.1038/bjc.2012.4. Epub 2012 Feb 7. PMID 22315052
- [Background] Klinkhammer-Schalke M, Koller M, Ehret C, Steinger B, Ernst B, Wyatt JC, Hofstadter F, Lorenz W; Regensburg QoL Study Group. Implementing a system of quality-of-life diagnosis and therapy for breast cancer patients: results of an exploratory trial as a prerequisite for a subsequent RCT. Br J Cancer. 2008 Aug 5;99(3):415-22. doi: 10.1038/sj.bjc.6604505. PMID 18665187
- [Background] Klinkhammer-Schalke M, Koller M, Wyatt JC, Steinger B, Ehret C, Ernst B, Hofstadter F, Lorenz W. Quality of life diagnosis and therapy as complex intervention for improvement of health in breast cancer patients: delineating the conceptual, methodological, and logistic requirements (modeling). Langenbecks Arch Surg. 2008 Jan;393(1):1-12. doi: 10.1007/s00423-007-0210-5. Epub 2007 Jul 28. PMID 17661076
- [Derived] Klinkhammer-Schalke M, Steinger B, Koller M, Zeman F, Furst A, Gumpp J, Obermaier R, Piso P, Lindberg-Scharf P; Regensburg QoL Study Group. Diagnosing deficits in quality of life and providing tailored therapeutic options: Results of a randomised trial in 220 patients with colorectal cancer. Eur J Cancer. 2020 May;130:102-113. doi: 10.1016/j.ejca.2020.01.025. Epub 2020 Mar 13. PMID 32179445
- [Derived] Klinkhammer-Schalke M, Lindberg P, Koller M, Wyatt JC, Hofstadter F, Lorenz W, Steinger B. Direct improvement of quality of life in colorectal cancer patients using a tailored pathway with quality of life diagnosis and therapy (DIQOL): study protocol for a randomised controlled trial. Trials. 2015 Oct 14;16:460. doi: 10.1186/s13063-015-0972-y. PMID 26467994